CLINICAL TRIAL: NCT03343899
Title: Identification of Genotype-related Molecular Targets in the Vitamin D Pathway for Personalized Pharmacological Treatments of the Spinal Disc Diseases
Brief Title: Genotype-related Molecular Targets in the Vitamin D Pathway for Spinal Disc Diseases
Acronym: GenVDisc
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: GenVDisc
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Intervertebral Disk Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of our study will be to analyze the interplay between particular VDR variants and its ligand in cells obtained from intervertebral disc and cartilage endplate and their action on cell proliferation and phenotype maintenance. The identification of novel molecular targets in the vitamin D pathway, potentially promoting pathological alterations of the tissues involved in spinal disc diseases, will allow to develop innovative and more personalized preventive and pharmacological/nutritional therapies.

ELIGIBILITY:
Inclusion Criteria:

patients with spinal disc diseases

* males and females
* 18≤age ≤ 70 years old
* Italian white
* patients with spinal disc diseases that will be surgically treated

Exclusion criteria:

- age < 18 or > 70 years old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with spinal disc diseases
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2016-02-17 (Actual); Primary Completion 2018-02-17 (Estimated); Study Completion 2019-02-17 (Estimated)

PRIMARY OUTCOMES:
Phenotype and genotype characterization | 1 year
  To evaluate structural alterations of the intervertebral disc and of the cartilage endplate in patients with spinal disc diseases related to functional FokI polymorphism in the vitamin D receptor (VDR) gene.

SECONDARY OUTCOMES:
Disc cell functional response genotype-based | 2 years
  To characterize cells obtained from different disc tissues (nucleus pulposus, annulus fibrosus, cartilage endplate) and to evaluate their VDR FokI genotype-related response to vitamin D treatment, regulating the cell proliferation and phenotype.

CONTACTS AND LOCATIONS:
Locations (1):
- Alessandra Colombini, Milan, Italy